CLINICAL TRIAL: NCT01347281
Title: Non Invasive Imaging of [18F]HX4 With Positron-Emission-Tomography (PET) in Head and Neck Cancer.
Brief Title: PET With [18F]HX4 in Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-12-23/03-intern-6470; 2011-001812-80 (EudraCT Number)
Record Dates: First submitted 2011-05-03; First posted 2011-05-04 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Cancer of the Head and Neck
Keywords: Cancer of the Head and Neck; [18F]HX4; hypoxia; PET; phase II trial
MeSH Terms: conditions — Head and Neck Neoplasms; Hypoxia | interventions — 3-fluoro-2-(4-((2-nitro-1H-imidazol-1-yl)methyl)-1H-1,2,3-triazol-1-yl)propan-1-ol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- [18F]HX4 PET (Experimental): Injection of [18F]HX4
  Interventions: Procedure: Injection of [18F]HX4

INTERVENTIONS:
Procedure: Injection of [18F]HX4 — Injection of [18F]HX4 before treatment (baseline) and after radiotherapy with 20 +/-4 Gy:
  [18F]HX4 PET scans; 444 MBq (12 mCi) [18F]HX4 administrated via a bolus IV injection. Image acquisition: static scan at 240 min p.i.
  Venous blood sampling: before injection of [18F]HX4 (blood hypoxia markers) Follow-up (3 months after treatment): [18F]FDG PET in treatment position

SUMMARY:
The aim of this study is to (i) Determine if tumor hypoxia can be accurately visualised with [18F] HX4 PET imaging in head and neck tumors (ii) correlate the [18F] HX4 PET images with blood and tissue markers and (iii) investigate the quality and optimal timing of [18F] HX4 PET imaging (iv) compare [18F] HX4 PET uptake with [18F] FDG PET uptake before and after treatment.

DETAILED DESCRIPTION:
Tumor hypoxia is the situation where tumor cells are or have been deprived of oxygen. Hypoxic tumor cells are usually more resistant to radiotherapy and chemotherapy and more likely to develop metastasis. In head and neck cancer, tumor hypoxia is known to be an important prognostic factor for long term survival. [18F]HX4 is being developed as a diagnostic radiopharmaceutical for PET imaging to find a marker for hypoxia that can be used in standard clinical practice. Current hypoxia tracers lack reliable image quality and kinetics. Because of the short half life and clearance, we expect that [18F]HX4 will have a higher tumor to background ratio than current nitro-imidazole hypoxia markers such as [18F]-misonidazole. The clinical use of a reliable, non-invasive and easy to use hypoxia imaging agent could allow selection of patients most likely to benefit from hypoxia modifying therapies.

Included are eligible patients with head and neck squamous cell carcinoma (T2, T3, T4, any N, M0) with tumor diameter ≥ 2,5 cm of the oral cavity, oropharynx, hypopharynx or larynx, planned to be treated with curative primary radiation treatment (+/- concurrent chemotherapy). Before treatment a standard planning [18F]FDG PET-CT will be performed, a blood sample is drawn and baseline [18F]HX4 PET scans will be performed. 18F-HX4 scans will be repeated after radiotherapy treatment with 20 +/- 4 Gy (approximately two weeks). Three months after the end of treatment a [18F]FDG PET scan will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed HNSSC of the oral cavity, oropharynx, hypopharynx, larynx, T2-T3-T4, any N, M0
* Tumor diameter ≥ 2,5 cm
* WHO performance status 0 to 2
* Scheduled for primary curative (concurrent chemo-) radiotherapy
* No previous surgery to the head and neck
* No previous radiation to the head and neck
* Adequate renal function (calculated creatinine clearance at least 60 ml/min).
* The patient is willing and capable to comply with study procedures
* 18 years or older
* Have given written informed consent before patient registration

Exclusion Criteria:

* No recent (< 3 months) myocardial infarction
* No Uncontrolled infectious disease
* Not pregnant or breast feeding and willing to take adequate contraceptive measures during the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-12; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Visualisation of tumor hypoxia with [18F] HX4 PET imaging | 2 years
  Visualisation of tumor hypoxia with [18F] HX4 PET imaging

SECONDARY OUTCOMES:
Observe spatial and temporal stability of [18F] HX4 PET images | 2 years
Correlation of [18F] HX4 with local tumor recurrence and survivalG PET | 2 years
Image quality of [18F] HX4-PET at different time points | 2 years
Kinetic analysis of HX4 | 2 years
Correlation of hypoxia imaging with blood hypoxia markers | 2 years
Correlation of hypoxia imaging with tumor tissue biomarkers | 2 years
Spatial correlation of [18F] HX4-PET with [18F] FDG PET pre-treatment | 2 years
Spatial correlation of [18F] HX4-PET with [18F] FDG PET three months after treatment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Philppe Lambin, Prof. Dr., Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- Maastricht Radiation Oncology (MAASTRO clinic), Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided